CLINICAL TRIAL: NCT01618604
Title: Quantitative Sensory Testing in Context With Conditioned Pain Modulation (CPM)
Brief Title: QST in Context With Conditioned Pain Modulation
Acronym: CPM
Status: Completed | Type: Observational
Sponsor: Ruhr University of Bochum (Other)
Responsible Party: Principal Investigator, Christoph Maier, Prof. Dr., Head of the Dep. of Pain Management, Ruhr University of Bochum
Other Study IDs: CPM2012
Record Dates: First submitted 2012-06-11; First posted 2012-06-13 (Estimated); Last update posted 2013-01-03 (Estimated); Status verified 2012-12

CONDITIONS: Healthy
Keywords: Conditioned Pain Modulation; Quantitative Sensory Testing; duration; correlation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Healthy: 26 healthy voluntary probands
  Interventions: Procedure: Quantitative Sensory Testing; Procedure: Conditioned Pain Modulation; Procedure: Repetition of four QST parameters

INTERVENTIONS:
Procedure: Quantitative Sensory Testing — following the standardized protocol of DFNS
  Other Names: QST
Procedure: Conditioned Pain Modulation — test stimulus by hot thermode conditioned stimulus by cold water bath
  Other Names: CPM; DNIC; Diffuse Noxious Inhibitory Controls
Procedure: Repetition of four QST parameters — * warm detection threshold (WDT)
  * cold detection threshold (CDT)
  * mechanical detection threshold (MDT)
  * mechanical pain threshold (MPT)
  Other Names: WDT; CDT; MDT; MPT; Quantitative Sensory Testing

SUMMARY:
Conditioned Pain Modulation (CPM) is a phenomenon which isn't examined enough. Many factors of influence such as gender, age and psyche are already known - but the duration of such effects, their reliability and the correlation between standardized Quantitative Sensory Testing (QST) and CPM is still unknown.

In this study the investigators expect to find parameters in QST that correlate with the efficacy of Conditioned Pain Modulation. Knowing factors that indicate high or low potential CPM could help finding patients-at-risk and adapting their therapy.

DETAILED DESCRIPTION:
Conditioned Pain Modulation was firstly found in rats by electrical stimulation of their spinal cord and called Diffuse Noxious Inhibitory Controls. In humans such experimental settings are impossible. That is why we need two noxious stimuli for provoking such an endogenous pain inhibition.

Before the CPM setting begins, we will investigate our 32 healthy probands by basic QST following the protocol of DFNS (German Research Network on Neuropathic Pain). This assessment helps us to create a sensory profile for every proband and to look for correlations between QST parameters and CPM efficacy. Then the CPM setting follows. In our experimental design we use a test stimulus (TS) on the dominant forearm by thermode (normally 45-47°C, depending on the pain rating, we need scores >NRS 60) and a conditioned stimulus (CS) on the other hand by cold water bath (10°C). Both stimuli must be rated on the numerical rating scale (NRS) 0-100 alone and in combination. A positive effect can be seen, if the difference between TS alone and TS in combination with CS is >0. To learn more about the duration of CPM effects we decided to repeat four QST parameters (cold detection threshold, warm detection threshold, mechanical detection threshold and mechanical pain threshold) within 30 minutes after finishing the CPM part to detect changes of time.

The whole study design will be repeated 24-72h hours later to increase the test-retest-reliability.

ELIGIBILITY:
Inclusion Criteria:

* healthy probands >18 years
* right-handedness
* informed consent
* no chronic pain
* no drugs (but oral contraceptives)
* no neurological diseases
* no psychiatric diseases

Exclusion Criteria:

* no informed consent
* language deficits
* left-handedness
* not enough pain intensity by thermode or cold water bath
* psychiatric disease, neurological diseases other chronic disease
* chronic pain syndromes
* pregnancy or lactation
* permanent drug use, drug use in the last 14 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy voluntary probands
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2012-05; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Maier, Prof. Dr. med, Study Director — University hospital Bergmannsheil department of pain management
Locations (1):
- Bergmannsheil, department for pain management, Bochum, North Rhine-Westphalia, Germany

REFERENCES:
- [Derived] Gehling J, Mainka T, Vollert J, Pogatzki-Zahn EM, Maier C, Enax-Krumova EK. Short-term test-retest-reliability of conditioned pain modulation using the cold-heat-pain method in healthy subjects and its correlation to parameters of standardized quantitative sensory testing. BMC Neurol. 2016 Aug 5;16:125. doi: 10.1186/s12883-016-0650-z. PMID 27495743